CLINICAL TRIAL: NCT03416426
Title: Residual Shunt After Patent Foramen Ovale Device Closure in Patients With Cryptogenic Stroke: Serial Bubble Contrast Transesophageal Echocardiography Data
Brief Title: Residual Shunt After Patent Foramen Ovale Device Closure in Patients With Cryptogenic Stroke
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Woong Chol Kang, Director of Cardiology, Gachon University Gil Medical Center
Other Study IDs: RSHUNT
Record Dates: First submitted 2018-01-11; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Patent Foramen Ovale; Closure; Foramen Ovale
Keywords: patent foramen ovale; PFO closure; residual shunt; bubble contrast transesophageal echocardiography
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- patients undergone PFO closure: patients with ischemic stroke and PFO documented by bubble contrast TEE with no other identifiable cause of the ischemic event who undergone PFO closure using Amplatzer® PFO occluder or Gore® Septal Occluder
  Interventions: Device: Amplatzer® PFO occluder or Gore® Septal Occluder

INTERVENTIONS:
Device: Amplatzer® PFO occluder or Gore® Septal Occluder — The closure procedure was performed under general anesthesia. After achieving femoral venous access, the PFO was crossed with a 5F multipurpose catheter, which was advanced into the left upper pulmonary vein and then exchanged over a 0.035 inch J-tipped stiff guidewire for an 8F or 9F guiding sheath. Procedural anticoagulation was initiated with 5000 units of intravenous heparin. After then additional heparin was administrated throughout procedure to maintain an activated clotting time of ≥250 seconds. Device size was selected based on TEE measurements of the distance between the PFO and the aortic root.

SUMMARY:
Among consecutive 47 cryptogenic stroke patients who underwent PFO closure, a serial follow-up bubble contrast TEE at 3 and 9 months after the index procedure was completed in 38 patients (81%, 46±10 years, 19 men). To evaluate the efficacy of PFO closure, the incidence of any- and significant residual shunt (≥moderate) was assessed.

DETAILED DESCRIPTION:
The current investigation analyzed the date from the Gachon University Gil Medical Center PFO registry. Between March 2014 to February 2017, all consecutive 47 patients with ischemic stroke and PFO documented by bubble contrast with no other identifiable cause of the ischemic event, such as, carotid or intracranial artery stenosis, atrial fibrillation, and thrombus, or atheromatous plaque at the aortic arch (i.e. CS), were analyzed. PFO closure was determined according to the heart-brain team's discretion (the team consisted of an interventional cardiologist, an echocardiographer cardiologist, a neurologist, and a radiologist) based on clinical data, echocardiographic findings, and patients' preference. The Gore® Septal Occluder (WL Gore & Associates, Inc., Newark, DE, USA) (n=19) and the Amplatzer® PFO occluder (St. Jude Medical, Inc. St.Paul, MN, USA) (n=19) and were used. The Occlutec® PFO occluder was used in one patient who were excluded from the analysis. The Institutional Review Board of Gachon University Gil Medical Center approved this study and all patients provided written informed consent prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

patients with cryptogenic stroke and PFO documented by bubble contrast TEE

Exclusion Criteria:

patients with other identifiable cause of the ischemic event such as, carotid or intracranial artery stenosis, atrial fibrillation, and thrombus, or atheromatous plaque at the aortic arch

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive 47 patients with ischemic stroke and PFO documented by BCTEE with no other identifiable cause of the ischemic event, such as, carotid or intracranial artery stenosis, atrial fibrillation, and thrombus, or atheromatous plaque at the aortic arch (i.e. CS), were analyzed. PFO closure was determined according to the heart-brain team's discretion (the team consisted of an interventional cardiologist, an echocardiographer cardiologist, a neurologist, and a radiologist) based on clinical data, echocardiographic findings, and patients' preference.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Residual shunt rate at 9 months | 9-month follow-up bubble contrast TEE
  Incidence of significant residual shunt (≥moderate) was assessed.

SECONDARY OUTCOMES:
Residual shunt rate at 3 months | 3-month follow-up bubble contrast TEE
  Incidence of significant residual shunt (≥moderate) was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Woong Chol Kang, MD, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No